CLINICAL TRIAL: NCT04893317
Title: Cryoablation for Monomorphic Ventricular Tachycardia
Brief Title: Cryoablation for Monomorphic Ventricular Tachycardia (CryoCure-VT)
Acronym: CryoCure-VT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adagio Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-098
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Monomorphic Ventricular Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation in the ventricle with the Adagio VT cryoablation system (Experimental): all study subjects will receive an ablation procedure using the Adagio Medical VT Cryoablation System
  Interventions: Device: Ablation in the ventricles with the Adagio Medical VT Cryoablation System

INTERVENTIONS:
Device: Ablation in the ventricles with the Adagio Medical VT Cryoablation System — The Adagio Medical VT Cryoablation System is indicated for the treatment of monomorphic ventricular tachycardia by ablation of arrhythmogenic tissue that drives and maintains these arrhythmias

SUMMARY:
A prospective, single-arm, multi-center, pre-market, clinical study designed to provide safety and performance data regarding the use of the Adagio Medical VT Cryoablation System in the treatment of ventricular tachycardia.

DETAILED DESCRIPTION:
Study subjects will include patients who experience recurrent monomorphic VT and are scheduled for an endocardial VT ablation. Study subjects have or will have an Implantable Cardioverter Defibrillator (ICD) prior to hospital discharge following the cryoablation procedure.

A VT ablation procedure is performed by finding the abnormal ventricular heart tissue that is causing the VT and applying energy with an ablation catheter to the area. The goal is to apply energy to create a scar or destroy the tissue that causes the VT, such that VT is no longer present or inducible.

ELIGIBILITY:
Inclusion Criteria:

IC 1 Male or female the ages of ≥ 18 years

IC 2 Eligible for a catheter ablation due to Ischemic and/or non-ischemic recurrent symptomatic sustained monomorphic Ventricular Tachycardia also defined as having a similar QRS configuration from beat to beat.

IC 3 Has or will be receiving an ICD prior to hospital discharge post procedure.

IC 4 Refractory to at least one AAD (Refractory is defined as an AAD not able to treat the arrhythmia satisfactorily or induces unwanted side effects).

IC 5 Subject has LVEF > 20%, confirmed by echo or comparable technique in the previous 3 months or during baseline evaluation

IC 6 Willingness, ability, and commitment to participate in baseline and follow-up evaluations for the full length of the study

IC 7 Willingness and ability to give an informed consent

Exclusion Criteria:

EC 1 Any known objective contraindication to ventricular tachycardia ablation, TEE, or anticoagulation, including but not limited to the identification of any cardiac thrombus or evidence of sepsis

EC 2 Any duration of continuous arrythmia that is not monomorphic ventricular tachycardia. Multiple monomorphic tachycardia is acceptable, but polymorphic VT is not.

EC 3 Any VT ablation within 4 weeks prior to enrollment

EC 4 More than one prior (>4 weeks) Ventricular Tachycardia ablation or prior surgical treatment for ventricular tachycardia

EC 5 Ventricular tachycardia secondary to electrolyte imbalance, active thyroid disease, or any other reversible or non-cardiac cause

EC 6 Structural heart disease as described below:

1. Class IV heart failure
2. Aortic aneurysm
3. Previous cardiac surgery or percutaneous coronary intervention within 60 days prior to the procedure
4. Interatrial baffle, closure device, patch, or PFO occlusion device
5. IVC filter
6. Coronary artery bypass graft (CABG) procedure within six (6) months prior to the ablation procedure
7. Severe Mitral or Aortic insufficiency or stenosis based on most recent TTE
8. Cardiac myxoma
9. Significant congenital anomaly
10. Recent Myocardial Infarct (MI) or unstable angina, within 60 days prior to the ablation procedure
11. Mechanical aortic or mitral valve

EC 7 Any previous history of cryoglobulinemia

EC 8 History of blood clotting or bleeding disease

EC 9 Any prior history of documented cerebral vascular accident (CVA), TIA or systemic embolism (excluding a post-operative Deep Vein Thrombosis, DVT), within 6 months prior to the ablation procedure.

EC 10 Breastfeeding, pregnant, or anticipated pregnancy during study follow-up

EC 11 Current enrollment in any other study protocol where testing or results from that study may interfere with the procedure or outcome measurements for this study

EC 12 Any other condition that, in the judgment of the investigator, makes the patient a poor candidate for this procedure, the study or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, candidate for heart transplantation, patient with ventricular assist device, or terminal illness with a life expectancy less than 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint for Safety | during and 30 days post cryoablation procedure
  An analysis of the proportion of subjects who are free from definite or probable device/procedure related Major Adverse Events (MAEs) that occur during or within 30 days following the cryoablation procedure
Primary Endpoint for Clinical Performance | 6 month post cryoablation procedure
  an analysis of the proportion of patients receiving a single cryoablation procedure with freedom from ventricular tachycardia lasting longer than 30 seconds or appropriate ICD intervention until the end of the 6 month follow up period.
Primary Endpoint for Procedure Performance | at the end of the cryoablation procedure
  an analysis of the proportion of subjects with non-inducible clinical monomorphic VT at the conclusion of the initial cryoablation procedure

SECONDARY OUTCOMES:
Safety - freedom from procedure or device related SAE | 12 months post cryoablation procedure
  The proportion of study subjects with probable or definite device or procedure related serious adverse events (SAEs) including MAEs as described above, or serious adverse device effects (SADEs) between 30-days up to 12 months post-procedure.
Performance - non-inducible sustained monomorphic VT | at the end of the cryoablation procedure
  The proportion of study subjects with non-inducible sustained monomorphic VT at the end of the ablation procedure
Performance - freedom from VT at 12-M off AADs | 12 months post cryoablation procedure
  The proportion of study subjects with freedom from Ventricular Tachycardia lasting longer than 30 seconds at 12 months without the use of anti-arrhythmic drugs (AADs)
Performance - freedom from VT at 12-M on previously failed AADs | 12 months post cryoablation procedure
  The proportion of study subjects with freedom from Ventricular Tachycardia lasting longer than 30 seconds at 12 months with previously failed anti-arrhythmic drugs (AADs)
Performance - VT burden | 6 and 12 months post cryoablation procedure
  Reduction of VT burden at 6 and 12 months
Descriptive Statistical Outcome - fluoroscopy time | at the end of the cryoablation procedure
  Procedure fluoroscopy time
Descriptive Statistical Outcome - ablation time | at the end of the cryoablation procedure
  Total ablation time
Descriptive Statistical Outcome - procedure time | at the end of the cryoablation procedure
  Total ablation time
Descriptive Statistical Outcome - cryoablation lesions | at the end of the cryoablation procedure
  Number and location of cryoablation lesions
Descriptive Statistical Outcome - inducible VTs | at the end of the cryoablation procedure
  Number of inducible clinical VTs before and after cryoablation
Descriptive Statistical Outcome - ICD shocks | 12 months post cryoablation procedure
  Number of appropriate and inappropriate ICD therapies (shocks and pacing) in the follow up period
Descriptive Statistical Outcome - ablation strategies | at the end of the cryoablation procedure
  Mapping and ablation strategies utilized during the ablation procedure
Descriptive Statistical Outcome - Hospitalization | 12 months post cryoablation procedure
  Freedom from cardiovascular (CV) hospitalizations or CV-related ER visits through 12 months
Descriptive Statistical Outcome - AADs use | 12 months post cryoablation procedure
  Recording of the use of AADs in the follow up period

CONTACTS AND LOCATIONS:
Locations (7):
- Onze Lieve Vrouwziekenhuis, Aalst, Belgium
- Canada (2):
  - McGill University Health Centre, Montreal
  - Montreal Hear Institute, Montreal
- Nemocnice na Homolce, Prague, Czechia
- CHU-Bordeaux, Pôle cardio-thoracique, Hôpital Haut-Lévêque, Bordeaux, France
- Herzzentrum Leipzig Universitätsklinik für Kardiologie, Leipzig, Germany
- St Antonius Ziekenhuis, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verma A, Essebag V, Neuzil P, Dyrda K, Balt J, Dinov B, Darma A, Arya A, Sacher F, Reddy VY, Boersma L, Grigorov I, De Potter T. Cryocure-VT: the safety and effectiveness of ultra-low-temperature cryoablation of monomorphic ventricular tachycardia in patients with ischaemic and non-ischaemic cardiomyopathies. Europace. 2024 Mar 30;26(4):euae076. doi: 10.1093/europace/euae076. PMID 38582974
- [Derived] De Potter T, Balt JC, Boersma L, Sacher F, Neuzil P, Reddy V, Grigorov I, Verma A. First-in-Human Experience With Ultra-Low Temperature Cryoablation for Monomorphic Ventricular Tachycardia. JACC Clin Electrophysiol. 2023 May;9(5):686-691. doi: 10.1016/j.jacep.2022.11.017. Epub 2023 Jan 18. PMID 36752466